CLINICAL TRIAL: NCT06759194
Title: Holmium Laser Versus Bipolar Enucleation of the Prostate in Management of Benign Prostatic Hyperplasia Patients With Large Prostates: A Non-inferiority Prospective Randomized Clinical Trial
Brief Title: HoLEP vs BipolEP in Management of BPH Patients With Large Prostates
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mostafa Mohamed Atef Abdelaziz Mostafa, Lecturer of Urology, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HoLEP vs BipolEP
Record Dates: First submitted 2024-12-30; First posted 2025-01-06 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Benign Prostatic Hyperplasia
Keywords: Holmium Laser Enucleation of Prostate (HoLEP); Benign Prostatic Hyperplasia (BPH); Bipolar Enucleation of Prostate (BipolEP)
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Holmium Laser Enucleation of the Prostate (HoLEP) (Active Comparator): Half of the BPH patients with large prostate admitted to the study will undergo Holmium Laser Enucleation of the Prostate (HoLEP)
  Interventions: Procedure: Holmium Laser Enucleation of the Prostate
- Bipolar Enucleation of the Prostate (BipolEP) (Active Comparator): Half of the BPH patients with large prostate admitted to the study will undergo Bipolar Enucleation of the Prostate (BipolEP)
  Interventions: Procedure: Bipolar Enucleation of the Prostate

INTERVENTIONS:
Procedure: Holmium Laser Enucleation of the Prostate — Enucleation of the prostate gland using holmium laser energy
  Arms: Holmium Laser Enucleation of the Prostate (HoLEP)
Procedure: Bipolar Enucleation of the Prostate — Enucleation of the prostate gland using bipolar energy
  Arms: Bipolar Enucleation of the Prostate (BipolEP)

SUMMARY:
This is a non-inferiority prospective randomized comparative clinical trial aiming to prove the non-inferiority of bipolar enucleation of the prostate in comparison to holmium laser enucleation of the prostate in management of benign prostatic hyperplasia patients with large prostates and in turn its feasibility as an alternative procedure in hospitals with limited resources

DETAILED DESCRIPTION:
Benign prostatic hyperplasia (BPH) is a prevalent condition among older men. It is characterized by non-cancerous enlargement of the prostate gland often leading to urinary obstruction and significant morbidity. In case of failure of medical treatment, surgical intervention is often required especially in patients with larger prostates. Surgical options in such cases include Holmium Laser Enucleation of the Prostate (HoLEP) and Bipolar Enucleation of the Prostate (BipolEP). These modalities have emerged as promising relatively minimally invasive treatment options in patients with large prostates. HoLEP, utilizing laser technology to enucleate prostatic tissue, has been associated with reduced intraoperative blood loss, shorter catheterization time, and quicker recovery in comparison to open prostatectomy. Likewise, BipolEP, utilizing bipolar energy for enucleation, offers the advantage of reduced bleeding and shorter operative time. Both HoLEP and BipolEP have demonstrated efficacy in improving lower urinary tract symptoms (LUTS) and alleviating obstruction in BPH patients with large prostates, but the comparative efficacy and safety of both techniques remains highly debated. This study aims to compare the efficacy and safety of these two surgical modalities aiming to provide valuable insights that can enhance clinical decision-making and patient care in BPH management.

ELIGIBILITY:
Inclusion Criteria:

* Age >50 years
* Prostate volume >80 ml
* Failure of or noncompliance with medical treatment
* IPSS >15
* Qmax <15 ml/sec
* Urinary retention and fixed catheters with poor results on trial of voiding without catheter

Exclusion Criteria:

* Patients with active UTI
* Prostate cancer
* Bladder carcinoma
* Urethral stricture
* Neurogenic bladder disorders
* Redo cases

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in peak flow rate | At 6 months after the procedure (HoLEP or BipolEP)
  Treatment efficacy will be evaluated by comparing the change in peak flow rate (Qmax) on uroflowmetry between the two groups

SECONDARY OUTCOMES:
Complications | At 6 months after the procedure (HoLEP or BipolEP)
  Treatment safety will be evaluated by collecting and analyzing any reported complication within the first 6 postoperative months. Complications will be reported using the modified Clavien-Dindo classification system.

CONTACTS AND LOCATIONS:
Overall Officials: Mostafa M. Mostafa, M.D., Principal Investigator — Assiut University
Locations (1):
- Assiut University Urology Hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be made available to protect privacy of patients

REFERENCES:
- [Background] Becker B, Herrmann TRW, Gross AJ, Netsch C. Thulium vapoenucleation of the prostate versus holmium laser enucleation of the prostate for the treatment of large volume prostates: preliminary 6-month safety and efficacy results of a prospective randomized trial. World J Urol. 2018 Oct;36(10):1663-1671. doi: 10.1007/s00345-018-2321-8. Epub 2018 May 5. PMID 29730838
- [Background] Tan AH, Gilling PJ. Holmium laser prostatectomy: current techniques. Urology. 2002 Jul;60(1):152-6. doi: 10.1016/s0090-4295(02)01648-5. PMID 12100945
- [Background] Neill MG, Gilling PJ, Kennett KM, Frampton CM, Westenberg AM, Fraundorfer MR, Wilson LC. Randomized trial comparing holmium laser enucleation of prostate with plasmakinetic enucleation of prostate for treatment of benign prostatic hyperplasia. Urology. 2006 Nov;68(5):1020-4. doi: 10.1016/j.urology.2006.06.021. Epub 2006 Nov 7. PMID 17095078
- [Background] Shoma AM, Ghobrial FK, El-Tabey N, El-Hefnawy AS, El-Kappany HA. A randomized trial of holmium laser vs thulium laser vs bipolar enucleation of large prostate glands. BJU Int. 2023 Dec;132(6):686-695. doi: 10.1111/bju.16174. Epub 2023 Sep 28. PMID 37667842